CLINICAL TRIAL: NCT03266055
Title: Prebiotic Effects of Blueberry in Overweight/Obese Individuals: Potential Role of the Gut Microbiota in Alleviating the Metabolic Syndrome.
Brief Title: Effects of Blueberry on Gut Microbiota and Metabolic Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marie-Claude Vohl, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BLEUET 2017-135
Record Dates: First submitted 2017-07-06; First posted 2017-08-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gut Microbiota; Metabolic Syndrome
Keywords: Blueberry; Diet
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry powder (Experimental)
  Interventions: Dietary Supplement: 50 g of blueberry powder, taken daily for 8 weeks
- Blueberry placebo powder (Placebo Comparator)
  Interventions: Dietary Supplement: 50g of placebo blueberry powder, taken daily for 8 weeks

INTERVENTIONS:
Dietary Supplement: 50 g of blueberry powder, taken daily for 8 weeks — Subjects will consume blueberry powder during 8 weeks to test the possible effects of blueberries on gut microbiota composition and on metabolic syndrome parameters.
  Arms: Blueberry powder
Dietary Supplement: 50g of placebo blueberry powder, taken daily for 8 weeks — Subjects will consume blueberry placebo powder to test if there is a significant difference on the impact on gut microbiota composition and metabolic syndrome parameters between this treatment and the active treatment (blueberry powder).
  Arms: Blueberry placebo powder

SUMMARY:
There is growing evidence that nutritional intervention with dietary polyphenols can positively modulate the gut microbiota to improve cardiometabolic health. Whether the beneficial effects of blueberries on obesity and the metabolic syndrome can be linked to their potential impact on the gut microbiota and intestinal integrity remains speculative at this time. Moreover, the mechanisms of action underlying health benefits associated to blueberry consumption are still unknown. The investigators are thus proposing to combine the study of metagenomics, transcriptomics and metabolomics to test whether a prebiotic activity of highbush blueberries can play a role in the prevention of obesity-linked metabolic syndrome in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopause women in good health
* Caucasians
* At least one of the following : BMI between 25 and 40 kg/m2 or Waist circumference ≥ 80 cm for women and ≥ 94 cm for men
* At least one of the following : TG ≥ 1.35 mmol/L or fasting insulinemia ≥ 42 pmol/L

Exclusion Criteria:

* Metabolic disorders (hypertension, diabetes, hypercholesterolemia)
* Regular use of medication affecting study parameters
* Use of natural health product in the last 3 months
* Use of antibiotics in the last 3 months
* Nicotine users
* Allergy or intolerance for blueberries
* Blueberry taste aversion
* More than 2 alcohol drinks par day
* Particular dietary habits (vegetarism, gluten-free diet, cetogenic diet...)
* Weight change of more than 5% in the last 3 months
* Surgery in the last 3 months or planed during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma insulin/glucose of overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 12 months
Changes in plasma lipids/lipoproteins of overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 12 months

SECONDARY OUTCOMES:
Changes in gene expression in overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 3-6 months
Changes in metabolites concentration in overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 3-6 months
Changes in the gut microbiota composition in overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 3-6 months
Changes in blood pressure of overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 12 months
Changes in intestinal integrity of overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 12 months
Changes in inflammation biomarkers of overweight/obese men and women taking either blueberry powder or placebo blueberry powder | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Vohl, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

REFERENCES:
- [Derived] Rousseau M, Horne J, Guenard F, de Toro-Martin J, Garneau V, Guay V, Kearney M, Pilon G, Roy D, Couture P, Couillard C, Marette A, Vohl MC. An 8-week freeze-dried blueberry supplement impacts immune-related pathways: a randomized, double-blind placebo-controlled trial. Genes Nutr. 2021 May 17;16(1):7. doi: 10.1186/s12263-021-00688-2. PMID 34000994